CLINICAL TRIAL: NCT03041636
Title: Administration of Jakafi (Ruxolitinib) to Patients With Previously Untreated High-Risk Chronic Lymphocytic Leukemia (CLL)/Small Lymphocytic Lymphoma (SLL): A Phase II Clinical Trial
Brief Title: Ruxolitinib Phosphate in Treating Patients With Previously Untreated Chronic Lymphocytic Leukemia/Small Lymphocytic Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2015-0570; NCI-2017-00478 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2015-0570 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2017-02-01; First posted 2017-02-03 (Estimated); Results first posted 2021-04-21 (Actual); Last update posted 2021-04-21 (Actual); Status verified 2021-03

CONDITIONS: Chronic Lymphocytic Leukemia/Small Lymphocytic Lymphoma; Untreated Chronic Lymphocytic Leukemia
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — ruxolitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (ruxolitinib phosphate) (Experimental): Patients receive ruxolitinib phosphate PO BID. Treatment continues for up to 3 years in the absence of disease progression or unacceptable toxicity. Treatment beyond 3 years may be permitted after discussion with the principal investigator.
  Interventions: Drug: Ruxolitinib; Drug: Ruxolitinib Phosphate

INTERVENTIONS:
Drug: Ruxolitinib — Given PO
  Other Names: INCB-18424; INCB18424; Oral JAK Inhibitor INCB18424
Drug: Ruxolitinib Phosphate — Given PO
  Other Names: INCB-18424 Phosphate; Jakafi

SUMMARY:
This phase II trial studies how well ruxolitinib phosphate works in treating patients with previously untreated chronic lymphocytic leukemia/small lymphocytic lymphoma. Ruxolitinib phosphate may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the effect of ruxolitinib phosphate (ruxolitinib) in patients with high-risk chronic lymphocytic leukemia (CLL)/small lymphocytic lymphoma (SLL) who do not require anti-neoplastic therapy according to the International Workshop on Chronic Lymphocytic Leukemia (IWCLL) 2008 recommendations and were either previously untreated or treated with Ibrutinib for less than 3 months and were deemed Ibrutinib intolerant:

Ia. On disease burden. Ib. The rate of complete response (CR) and partial response (PR) as assessed by the IWCLL 2008 response criteria.

SECONDARY OBJECTIVES:

I. To evaluate the time to next treatment of high-risk CLL/SLL who do not require anti-neoplastic therapy according to the IWCLL 2008 recommendations.

OUTLINE:

Patients receive ruxolitinib phosphate orally (PO) twice daily (BID). Treatment continues for up to 3 years in the absence of disease progression or unacceptable toxicity. Treatment beyond 3 years may be permitted after discussion with the principal investigator.

After completion of study treatment, patients are followed up at 30 days.

ELIGIBILITY:
Inclusion:

1. Subjects who are able to understand and sign an informed consent document.
2. Subjects 18 years of age or older.
3. Subjects must be diagnosed with CLL/SLL and do not meet the IWCLL criteria for treatment
4. Patients should be previously untreated or have only been treated with single agent ibrutinib therapy for a period of < 3 months and were deemed ibrutinib intolerant.
5. Patients whose expected time to CLL/SLL treatment, according to our nomogram posted on the leukemia protocol priority list, is four years of less.
6. Subjects with hemoglobin values at the screening visit equal to or greater than 12.0 g/dL.
7. Subjects with a platelet count of at least 100 x10^9 at the screening visit.
8. Subjects with an absolute neutrophil count (ANC) of equal to or higher than 0.5 x10^9 at the screening visit.
9. Subject who are willing to undergo a bone marrow aspiration and biopsy and CT scan for disease burden assessment.
10. Patient who are capable to return to MD Anderson Cancer Center (MDACC) for follow-up
11. Subjects with an Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1 or 2
12. Patient must be capable of swallowing the Ruxolotinib capsules (tablets).

Exclusion:

1. Females who are pregnant or are currently breastfeeding.
2. Subjects of childbearing potential who are unwilling to take appropriate precautions (throughout the study from screening including 30 days after discontinuation of the study drug) to avoid becoming pregnant or fathering a child. A) Females of non-childbearing potential are defined as women who (a) are equal to or greater than 55 years of age with history of amenorrhea for 1 year, OR (b) are surgically sterile for at least 3 months. B) For females of childbearing potential, or for males, appropriate precautions are those that are at least 99% effective in preventing the occurrence of pregnancy. These methods should be communicated to the subjects and their understanding confirmed: a) Double barrier methods; b) Condom with spermicide in conjunction with use of an intrauterine device (IUD); c) Condom with spermicide in conjunction with use of a diaphragm; d) Oral, injectable, or implanted contraceptives; e) Tubal ligation or vasectomy (surgical sterilization)
3. Subjects with recent history of inadequate bone marrow reserve as demonstrated by previous transfusions except for acute blood loss (e.g. surgery) in the month prior to screening.
4. Subjects with inadequate liver or renal function at screening and baseline visits: A) Alanine aminotransferase (ALT) > 2.5x Upper limit of normal (ULN). B) Modification of Diet in Renal Disease (MDRD) calculated GFR < 30 mL/min
5. Subjects with active uncontrolled infection or who are HIV positive (Subjects with acute infections requiring treatment should delay screening/enrollment until the course of therapy has been completed and the event is considered controlled).
6. Subjects with a history of or a current malignancy except for treated basal or squamous carcinomas of the skin completely resected.
7. Subjects with clinically significant uncontrolled cardiac disease.
8. Subjects being treated concurrently with any prohibited medications, including investigational medication, rifampin, St. John's wort, and potent CYP3A4 inhibitors (excluding ketoconazole) unless continuation of such medications are determined by the investigator to be in the best interest of the patient. Refer to protocol section 2.2.12 for more details.
9. Subjects who have previously received JAK inhibitor therapy
10. Subjects with active alcohol or drug addiction that would interfere with their ability to comply with the study requirements.
11. Subjects with any concurrent condition that, in the Investigator's opinion, would jeopardize the safety of the subject or compliance with the protocol.
12. Subjects who have unknown transfusion history.
13. Patients who cannot comply with the study requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2017-03-08 (Actual); Primary Completion 2020-04-29 (Actual); Study Completion 2020-04-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Zeev Estrov, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: March 2017 to June 2019
Groups:
- Treatment (Ruxolitinib Phosphate): Patients receive ruxolitinib phosphate PO twice a daily (BID). Treatment continues for up to 3 years in the absence of disease progression or unacceptable toxicity. Treatment beyond 3 years may be permitted after discussion with the principal investigator.
  Ruxolitinib: Given PO
  Ruxolitinib Phosphate: Given PO
Period: Overall Study
Arm/Group | Treatment (Ruxolitinib Phosphate)
Started | 1
Completed | 1
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Ruxolitinib Phosphate)
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 1
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 1

OUTCOME MEASURES:

1. Primary Outcome: Participants With a Clinical Response
Description: Clinical response will be assessed based on physical examination, complete blood count (CBC), a bone marrow aspiration, a whole body CT scan to be done at screening and 6 + 2 months in accordance with the International Workshop on Chronic Lymphocytic Leukemia (IWCLL) guidelines (Hallek et al., 2008)
Time Frame: Up to 6 months after initiation of therapy
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Ruxolitinib Phosphate)
Number analyzed (Participants) | 1
Participants | 0

2. Primary Outcome: Number of Participants With Change of Tumor Burden
Description: Tumor burden will be assessed by bone marrow aspiration, whole body CT scan at screening and 6 months.
Time Frame: 6 months after initiation of therapy
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Ruxolitinib Phosphate)
Number analyzed (Participants) | 1
Participants | 0

3. Primary Outcome: Participants With a Response
Description: Response Rate is Complete Response (CR) or Partial Response (PR). CR is absence of Lymphadenopathy, Hepatomegaly or Splenomegaly, lymphocytes < 4000/ul, normocellular, <30% lymphocytes, no B-lymphoid nodules, Platelets > 100,000/ul, hemoglobin >11.0 g/dl and Neutrophils >1500/ul.
  PR is >/= 50% decrease in lymphadenopathy, hepatomegaly, splenomegaly and Blood Lymphocytes from baseline, 50% reduction in marrow infiltrate or B-lymphoid nodules. Platelet count > 100,000/ul, Hemoglobin > 11 g/dl and Neutrophils >1500/ul or increase >/= 50% of all over base.
Time Frame: Up to 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Ruxolitinib Phosphate)
Number analyzed (Participants) | 1
Participants | 0

4. Primary Outcome: Time to Next Treatment
Description: Number of months to subsequent therapy per patient.
Time Frame: Up to 30 days
Measure: Number; unit: Months
Arm/Group | Treatment (Ruxolitinib Phosphate)
Number analyzed (Participants) | 1
Months | 0

ADVERSE EVENTS:
Time Frame: Up to 3 years
Arm/Group | Treatment (Ruxolitinib Phosphate)
All-Cause Mortality (participants affected / at risk) | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 1/1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Ruxolitinib Phosphate) (N=1)
Skin Infection (Infections and infestations) | 1 (1)
Upper Respiratory Infection (Infections and infestations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-03-02): https://cdn.clinicaltrials.gov/large-docs/36/NCT03041636/Prot_SAP_000.pdf